CLINICAL TRIAL: NCT00885846
Title: A Pilot Study: The Effects of Qigong Therapy on Type 2 Diabetic Patients
Brief Title: Effects of Qigong on Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bastyr University (Other)
Collaborators: Seattle Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H77B11
Record Dates: First submitted 2009-02-05; First posted 2009-04-22 (Estimated); Results first posted 2009-04-22 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Qigong; Breathing management; Glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (3):
- Qigong Therapy (Active Comparator)
  Interventions: Other: Qigong therapy
- PRT (Active Comparator)
  Interventions: Other: Progressive resistance training
- Control (No Intervention)

INTERVENTIONS:
Other: Qigong therapy — For 12 weeks, subjects in Qigong therapy group are to follow a disciplined regular practice, 3 times a week for about 30 minutes, including once a week with a certified instructor to lead and check the correctness of their practice.
  Arms: Qigong Therapy
Other: Progressive resistance training — For 12 weeks, subjects in the PRT group are to follow a disciplined regular practice, 3 times a week for about 30 minutes, including once a week with a certified instructor to lead and check the correctness of their practice.
  Arms: PRT

SUMMARY:
Qigong therapy is a subtle energy-based methodology for preventing and healing diseases that has been practiced with remarkable results in China for about five thousand years. Recently, preliminary studies showed that Qigong exercises improve insulin resistance and glucose metabolism in people with type 2 diabetes. These studies suggest that Qigong therapy might be an effective and valuable complementary modality for treating type 2 diabetes. Type 2 diabetes is a chronic disease marked by abnormally high levels of sugar in the blood. Diabetes is a serious disease, which, if not controlled, can be life threatening.

The purpose of this project is to conduct a randomized, controlled pilot clinical trial to compare the effectiveness of Qigong therapy to mild exercise and conventional treatment in type 2 diabetes and to identify biological and psychological characteristics associated with subjects' responses to Qigong therapy.

Aim 1: To compare the effects on blood sugar and hemoglobin A1c (HbA1c) level between a Qigong therapy group and non-treated control group as well as between Qigong group and a progressive resistance training (PRT) group before, during and after and 12-week intervention.

Hypothesis 1: Both Qigong therapy and PRT will help type 2 diabetic patients reduce blood sugar levels to different degrees through improving insulin resistance. But the levels of reduction of blood sugar will be greater by Qigong therapy than by PRT due to enhanced insulin secretion.

Aim 2: To compare the effects on fasting C-peptide and insulin levels between a Qigong therapy group, a PRT group and a non-treated control group before and after the intervention.

Hypothesis 2: Qigong therapy will increase the endogenous insulin and C-peptide levels by restoring the functions of the pancreas, while PRT will not alter either insulin or C-peptide levels.

Aim 3: To compare the effects of Qigong therapy and PRT on blood cortisol levels and psychological stress levels before, during and after the intervention.

Hypothesis 3: Perceived stress and depression will be improved by Qigong therapy to a greater extent than by PRT, and blood cortisol levels will be reduced to a greater extent with Qigong therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes defined as a glycohemoglobin between 7.5% and 10.5%, and fasting insulin level <40 (IU/ml).
* Must be controlling their diabetes with diet or may be taking oral medication for at least three months
* Age 18-65
* Ability to physically perform Qigong or low-intensity physical exercise
* Body Mass Index 18-40
* Have current primary care
* Willing to monitor blood glucose at least twice a day
* Willing to maintain a consistent diet during the study, and
* Sign informed consent

Exclusion Criteria:

* Significant kidney, liver or heart disease
* History of drug or alcohol abuse within the past 2 years
* Current or previous use of insulin
* Use of dietary supplements that affect blood glucose or insulin
* Current practice of Qigong (any style)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-06; Primary Completion 2008-01 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guan-Cheng Sun, PhD, Principal Investigator — Bastyr University; Jennifer C Lovejoy, PhD, Study Director — Bastyr University; Ryan Bradley, ND, Study Chair — Bastyr University
Locations (1):
- Bastyr University Research Center, Kenmore, Washington, United States

REFERENCES:
- [Background] Tsujiuchi T, Kumano H, Yoshiuchi K, He D, Tsujiuchi Y, Kuboki T, Suematsu H, Hirao K. The effect of Qi-gong relaxation exercise on the control of type 2 diabetes mellitus: a randomized controlled trial. Diabetes Care. 2002 Jan;25(1):241-2. doi: 10.2337/diacare.25.1.241. No abstract available. PMID 11772923
- [Background] Iwao M, Kajiyama S, Mori H, Oogaki K. Effects of qigong walking on diabetic patients: a pilot study. J Altern Complement Med. 1999 Aug;5(4):353-8. doi: 10.1089/acm.1999.5.353. PMID 10471015
- [Background] Xin L, Miller YD, Brown WJ. A qualitative review of the role of qigong in the management of diabetes. J Altern Complement Med. 2007 May;13(4):427-33. doi: 10.1089/acm.2006.6052. PMID 17532735
- [Derived] Sun GC, Lovejoy JC, Gillham S, Putiri A, Sasagawa M, Bradley R. Effects of Qigong on glucose control in type 2 diabetes: a randomized controlled pilot study. Diabetes Care. 2010 Jan;33(1):e8. doi: 10.2337/dc09-1543. No abstract available. PMID 20040671

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant recruitment for cohort 1: August 2007. Participant recruitment for cohort 2: February 2008. Place of recruitment: Bastyr University Research Institute.
Pre-assignment Details: The second cohort was necessary to achieve desired sample size.
Groups:
- Qigong Therapy: Participants practiced Qigong at least three times per week for 30 minute sessions, including once a week with a certified instructor, for 12 weeks.
- Progressive Resistance Training (PRT): Participants practiced PRT at least three times per week for 30 minute sessions, including once a week with a certified instructor, for 12 weeks.
- Non-treated Control: Participants were asked to maintain their conventional diabetes care for the duration of the study (12 weeks).
Period: Overall Study
Arm/Group | Qigong Therapy | Progressive Resistance Training (PRT) | Non-treated Control
Started | 11 (Cohort 1 = 5 Cohort 2 = 6) | 11 (Cohort 1 = 6 Cohort 2 = 5) | 10 (Cohort 1 = 4 Cohort 2 = 6)
Completed | 9 (Cohort 1 = 3 Cohort 2 = 6) | 6 (Cohort 1 = 1 Cohort 2 = 5) | 8 (Cohort 1 = 4 Cohort 2 = 6)
Not Completed | 2 | 5 | 2
Not completed — Withdrawal by Subject | 2 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Qigong Therapy | Progressive Resistance Training (PRT) | Non-treated Control | Total
Number analyzed (Participants) | 11 | 11 | 10 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0.0
  Between 18 and 65 years | 11 | 9 | 7 | 27.0
  >=65 years | 0 | 2 | 3 | 5.0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (7.5) | 52.8 (9.9) | 60.2 (6.3) | 56.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 6 | 19.0
  Male | 4 | 5 | 4 | 13.0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 10 | 32.0

OUTCOME MEASURES:

1. Secondary Outcome: Fasting C-peptide
Time Frame: weeks 0 and 12
Reporting Status: Not Posted

2. Secondary Outcome: Fasting Insulin
Time Frame: weeks 0 and 12
Reporting Status: Not Posted

3. Secondary Outcome: Perceived Stress Scale (PSS)
Time Frame: weeks 0 and 12
Reporting Status: Not Posted

4. Secondary Outcome: Beck's Depression Inventory (BDI)
Time Frame: weeks 0 and 12
Reporting Status: Not Posted

5. Secondary Outcome: HOMA-IR Index
Time Frame: weeks 0 and 12
Reporting Status: Not Posted

6. Secondary Outcome: Fasting Cortisol
Time Frame: Weeks 0 and 12
Reporting Status: Not Posted

7. Primary Outcome: Fasting Blood Glucose
Time Frame: Week 0 (baseline) and week 12 (final)
Population: Analysis performed per protocol. Participants excluded from analysis for changing or discontinuing medication during intervention.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Qigong Therapy | Progressive Resistance Training (PRT) | Non-treated Control
Number analyzed (Participants) | 7 | 5 | 8
mg/dL
  week 0 (baseline) | 184.9 (35.3) | 143.8 (35.0) | 156.4 (36.6)
  week 12 (final) | 161.9 (40.5) | 154.0 (44.7) | 168.4 (49.1)
Statistical Analysis 1: Comparison: Qigong Therapy vs Progressive Resistance Training (PRT) vs Non-treated Control; Power analysis suggested 27 participants, 9 in each group; Test type: Non-Inferiority or Equivalence — Regression analysis performed for equal variance at baseline; p = 0.664, Repeated ANOVA; degrees of freedom = 2

ADVERSE EVENTS:
Groups:
- Control: Wait list group; no activity at this arm. On list to start Qigong
Arm/Group | Qigong Therapy | Progressive Resistance Training | Control
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/10

LIMITATIONS AND CAVEATS:
Limitations to this study include high withdrawal rate from PRT group, especially during the first cohort. Also, participants from both Qigong and PRT group changed or discontinued medications. Consequently, their results were excluded from analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes